CLINICAL TRIAL: NCT04454814
Title: Postoperative Pain Incidence of Asymptomatic Mandibular Molar Teeth After Using Different Engine-driven Systems
Brief Title: Postoperative Pain After Root Canal Preparation Using Different Engine-driven Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Kandemir Demirci, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-6/15
Record Dates: First submitted 2020-06-26; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Asymptomatic Molar Teeth With Periapical Lesions
Keywords: one-visit root canal treatment,; engine-driven instruments,; asymptomatic molar teeth wtih periapical lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotary Engine-driven Instruments (Active Comparator): The instrumentation protocol with Protaper Universal rotary files was began with an S1 file with a brushing movement to the two thirds of the working length and then an SX file was introduced to the two thirds of the working length with a brushing movement Afterwards, S1, S2, F1, F2 files in mesial roots and F4 files in distal roots were used to the working length, respectively. Protaper F2 instrument was then used to complete the canal preparation in mesial roots and Protaper F4 instrument was used to complete the canal preparation in distal roots.
  Interventions: Other: Protaper Universal instruments
- Reciprocal Engine-driven Instruments (Active Comparator): The instrumentation of the root canal in the Reciproc Blue group began with a R25 instrument with a slow in-and-out pecking movement.According to the manufacturer instructions, a #10 K-file was inserted to the canal to check the canal is free to 1 mm beyond the prepared canal section. After each 3 pecks or when a resistance was encountered the instrument was pulled out of the canal. Afterward, the R25 instrument was inserted in to root canal until approximately two thirds of the working length.RB R25 instrument was then used to complete the canal preparation in mesial roots and RB R40 instrument was used to complete the canal preparation in distal roots.
  Interventions: Other: Reciproc Blue instruments

INTERVENTIONS:
Other: Protaper Universal instruments — Root canal treatment using Protaper Universal instruments
  Arms: Rotary Engine-driven Instruments
Other: Reciproc Blue instruments — Root canal treatment using Reciproc Blue instruments
  Arms: Reciprocal Engine-driven Instruments

SUMMARY:
A hundred twenty patients who had an asymptomatic mandibular molar teeth with periapical lesion were included. For each patient, teeth were prepared with Reciproc Blue or Protaper Universal instruments. Each tooth was obturated with gutta-percha and resin-based sealer using single cone technique for mesial roots and for distal roots single cone and cold lateral compaction technique. Root canal treatment was performed in a single visit. Postoperative pain was assessed as no, mild, moderate, or severe at 6, 12, 24, 48, 72 hours and 7 days after obturation.

DETAILED DESCRIPTION:
The aim of this study was to compare the effect of root canal preparation techniques on the occurrence and intensity of postoperative pain in patients with asymptomatic mandibular molar teeth with periapical lesions.A hundred twenty patients who had an asymptomatic mandibular molar teeth with periapical lesion were included. For each patient, teeth were prepared with Reciproc Blue or Protaper Universal instruments. Each tooth was obturated with gutta-percha and resin-based sealer using single cone technique for mesial roots and for distal roots single cone and cold lateral compaction technique. Root canal treatment was performed in a single visit. Postoperative pain was assessed as no, mild, moderate, or severe at 6, 12, 24, 48, 72 hours and 7 days after obturation.For the comparison of pain scores between the tested instrumentation systems, the Mann Whitney test was used. Differences between postoperative pain intencity for each instrumentation technique, at different time intervals, were assessed by the Friedman test. For the association of pain and an analgesic intake with gender, the chi-square test was performed. For the association of pain with age and an analgesic intake were calculated using Mann Whitney test. A P value < .05 or less was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients without systemic diseases
* Patients who had a mandibular first molar with asymptomatic periapical lesion without previous endodontic treatment with no sensitivity to percussion
* Patients who had no spontaneous pre-treatment pain
* Patients not having taken any analgesics, antibiotics or corticosteroids before the treatment visit,
* Patients who had no allergic reaction to NaOCl and no intolerance to nonsteroidal anti-inflammatory drugs.

Exclusion Criteria:

* Patients who had severe periodontal disease
* The teeth with previous endodontic treatment
* The teeth with root canal calcification, root resorption
* The teeth that could not be isolated with rubber dam or were not suitable for further restoration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative pain | 6-hour to 7-day
  Postoperative pain after 6, 12, 24, 48, 72 hours and 7 days after obturation was measured using a modified 4-grade visual analogue scale (VAS) ranging from 1(no pain), 2(mild pain), 3 (moderate pain/pain relieved by analgesics), to (4) severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Kandemir Demirci, Principal Investigator — Ege University Faculty of Dentistry; Seniha Miçooğulları Kurt, Study Chair — Ege University Faculty of Dentistry; Burcu Serefoglu, Study Chair — Ege University Faculty of Dentistry; Mehmet E Kaval, Study Chair — Ege University Faculty of Dentistry; Mehmet K Çalışkan, Study Chair — Ege University Faculty of Dentistry
Locations (1):
- Gözde Kandemir Demirci, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mollashahi NF, Saberi EA, Havaei SR, Sabeti M. Comparison of Postoperative Pain after Root Canal Preparation with Two Reciprocating and Rotary Single-File Systems: A Randomized Clinical Trial. Iran Endod J. 2017 Winter;12(1):15-19. doi: 10.22037/iej.2017.03. PMID 28179917
- [Background] Shokraneh A, Ajami M, Farhadi N, Hosseini M, Rohani B. Postoperative endodontic pain of three different instrumentation techniques in asymptomatic necrotic mandibular molars with periapical lesion: a prospective, randomized, double-blind clinical trial. Clin Oral Investig. 2017 Jan;21(1):413-418. doi: 10.1007/s00784-016-1807-2. Epub 2016 Apr 4. PMID 27041109
- [Result] Kherlakian D, Cunha RS, Ehrhardt IC, Zuolo ML, Kishen A, da Silveira Bueno CE. Comparison of the Incidence of Postoperative Pain after Using 2 Reciprocating Systems and a Continuous Rotary System: A Prospective Randomized Clinical Trial. J Endod. 2016 Feb;42(2):171-6. doi: 10.1016/j.joen.2015.10.011. Epub 2015 Nov 29. PMID 26614017
- [Result] Gambarini G, Sudani DA, Carlo SD, Pompa G, Pacifici A, Pacifici L, Testarelli L (2013) Incidence and intensivity of postoperative pain and periapical inflammation after endodontic treatment with two different instrumentation techniques. European Journal of Inflammation. 10, 99-103.